CLINICAL TRIAL: NCT00480246
Title: A Positron Emission Tomography (PET) Study to Assess the Degree of Dopamine-2 (D2) Receptor Occupancy in the Human Brain After Single Doses of BL-1020 or Perphenazine in Healthy Male Subjects Using [11C]Raclopride as PET Tracer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioLineRx, Ltd. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: BL- 1020.02
Record Dates: First submitted 2007-05-28; First posted 2007-05-30 (Estimated); Last update posted 2009-07-21 (Estimated); Status verified 2007-05

CONDITIONS: Healthy
Keywords: receptor oocupancy
MeSH Terms: interventions — perphenazine GABA ester; Perphenazine

INTERVENTIONS:
Drug: BL 1020
Drug: Perphenazine

SUMMARY:
This is a single dose, open-label, 2-panel (Parts A and B) PET study investigating the degree of occupancy of dopamine 2 receptors (D2_RO) in the human brain after single oral doses of BL-1020 or Perphenazine (Trilafon®, hereafter called Perphenazine) in healthy male subjects. In Part A the D2_RO is investigated for the study compound BL-1020 and in Part B the D2_RO of BL-1020 is compared to the D2_RO of Perphenazine, a reference compound.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed written informed consent agreement approved by the Independent Ethics Committee (IEC) after explanation of the nature and objectives of the study and prior to any study specific procedure.
2. Healthy male subjects between the age of 21 and 35 (inclusive).
3. Body Mass Index (BMI) (weight [kg] / (height [m] x height [m])) ≥ 18 and < 29 kg/m2.
4. Non-smokers or having refrained from smoking and other nicotine containing products for the last 1 month before dose administration.
5. Good health, based upon the results of medical history, physical examination, ECG (without clinically significant abnormalities) and laboratory profile of both blood and urine, including creatinine clearance, calculated using the Cockcroft-Gault formula (upper limit for eligibility 1.5 times the upper normal limit).
6. Normal blood pressure (systolic blood pressure ≥ 95 and ≤ 149 mmHg; diastolic blood pressure ≥ 55 and ≤ 89 mmHg) measured after 5 minutes rest in supine position.
7. Pulse rate of ≥ 45 and ≤ 95 beats/min measured after 5 minutes rest in supine position.
8. Able to communicate well with the investigator and able to comply with the requirements of the entire study.

Exclusion Criteria:

1. Intake of prescribed medication or Over the Counter (OTC) medication, including herbal remedies, minerals and vitamin preparations, within 14 days prior to dosing or scheduled to receive it during the study. Paracetamol is allowed, except for within 24 hours before each PET scan.
2. Demonstration of any active physical disease, acute or chronic.
3. Any gastrointestinal complaints within 7 days prior to dosing day.
4. Any condition which might interfere with the absorption of the investigational product, e.g. cholecystectomy (gall bladder removal, cholecystolithiasis).
5. Any relevant history of chronic or recurrent metabolic (e.g., diabetes), renal, hepatic, pulmonary, gastrointestinal (e.g., gastrointestinal disease, chronic gastritis or peptic ulcers), neurological (especially history of seizures disorders), endocrinological, immunological, psychiatric or cardiovascular disease, myopathies and bleeding tendency.
6. Positive test result for hepatitis B surface antigen (HBsAg), anti-Hepatitis C Virus (HCV) or Human Immunodeficiency Virus (HIV).
7. CYP2D6 genotype poor metabolizer.
8. Relevant drug hypersensitivity, asthma, urticaria or other severe allergic diathesis as well as ongoing hay fever.
9. Febrile or infectious illness within 7 days prior to the dosing day.
10. Participation in an investigational drug study within 3 months prior to the dosing day.
11. Donation of blood within 3 months prior to the dosing day.
12. History of alcoholism or more than moderate alcohol consumption (> 3 units of ethanol regularly per day or > 21 units regularly per week).
13. Consumption of alcohol within 48 hours prior to dose administration and/or positive alcohol breath test.
14. History of drug addiction or a positive drug urine screen for amphetamine, benzodiazepine, cannabis, cocaine, methadone or opiates.
15. Consumption of more than 5 cups of coffee or equivalent per day.
16. Consumption of xanthine-containing food or beverages, or grapefruit juice within 48 hours prior to dose administration.
17. Previous participation in a PET investigation.
18. Occupational exposure to significant ionizing radiation.
19. Having undergone any clinical procedure involving significant exposure to radiation (exceptions are e.g. dental X rays and common X-rays of chest or extremities), as judged by the investigator.
20. Suffers from claustrophobia.
21. Unsuitability for any other reason in the opinion of the investigator.

Ages: 21 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2007-05

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Wickström, Principal Investigator — Quintiles AB, Phase I Services
Locations (1):
- Quintiles Phase I facility, Uppsala, Sweden